CLINICAL TRIAL: NCT03108248
Title: Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis: Survival Benefit of Transarterial Chemoembolization in Combination With Irradiation Stent Placement
Brief Title: ISP-TACE Versus TACE for HCC With PVTT
Status: Completed | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Dr, Zhongda Hospital
Other Study IDs: ZhongdaHP
Record Dates: First submitted 2017-04-04; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: HCC; Portal Vein Tumor Thrombosis
Keywords: transarterial chemoembolization; stent; irradiation; survival; decompensation; tumor response
MeSH Terms: interventions — Ethiodized Oil; Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ISP-TACE group: During the study period, a total of 44 patients with HCC with PVTT underwent the irradiation stent placement and TACE were included in the ISP-TACE group.
  Interventions: Drug: ethiodized oil; doxorubicin;Gelfoam;
- TACE group: During the study period, a total of 82 patients with HCC with PVTT underwent TACE monotherapy were included in the ISP-TACE group.
  Interventions: Drug: ethiodized oil; doxorubicin;Gelfoam;; Device: stent; idoine-125

INTERVENTIONS:
Drug: ethiodized oil; doxorubicin;Gelfoam; — Conventional TACE was performed in both groups as follows. First, multiple angiographies were performed to detect the hepatic arterial anatomy and the possible feeding arteries of tumor, selective catheterization of the artery feeding the tumors was performed. A mixture of ethiodized oil was injected, followed by injection of Gelfoam particles.
Device: stent; idoine-125 — In the ISP-TACE group, stent placement was performed one week before TACE. Under fluoroscopic and ultrasonic guidance, the outer stent was firstly placed at the site of the obstructed portal vein, and a self-expandable nitinol stent was immediately followed through a same 10-F sheath.
  Groups: TACE group

SUMMARY:
For patients with advanced hepatocellular carcinoma (HCC) and portal vein tumor thrombosis (PVTT), the survival benefit of transarterial chemoembolization (TACE) remains modest. This study aimed to investigate whether TACE in combination with irradiation stent placement (ISP) could prolong the survival in patients with HCC and PVTT.

ELIGIBILITY:
Inclusion Criteria:

* (1) newly diagnosed HCC with type II or III PVTT, (2) Child-Pugh classification grade A or B, (3) Eastern Cooperative Oncology Group (ECOG) performance status score 0-2.

Exclusion Criteria:

* (1) type I or IV PVTT, (2) received sorafenib, systemic chemotherapy, or external radiotherapy during the treatment, (3) suffered from malignancy other than HCC, (4) with an incomplete data.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 2011 and December 2016, patients with HCC and PVTT underwent TACE combined with irradiation stent placement or TACE monotherapy as an initial treatment at the authors' center were retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2017-03-25 (Actual)

PRIMARY OUTCOMES:
survival | 0-6 years
  The overall survival (OS) was defined as the time from first treatment to death or the patient's last follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital,Southeast University, Nanjing, Jiangsu, China